CLINICAL TRIAL: NCT03771313
Title: Pharmacokinetic and Pharmacodynamic Analysis of Ceftaroline in Children and Adolescents With Cystic Fibrosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ceftaroline CF PK/PD_2017-2276
Record Dates: First submitted 2018-07-11; First posted 2018-12-11 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2024-11

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Ceftaroline

STUDY DESIGN:
Intervention Model Description: Open-label, single center, prospective study
Masking Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PK/PD (Other): Open-label prospective study with participants receiving treating physician-approved intravenous ceftaroline, dosed according to current recommendations. Blood samples collected at baseline, 1 hour, 1.5 hours, 3 hours, and 6 hours after infusion.
  Interventions: Drug: Ceftaroline

INTERVENTIONS:
Drug: Ceftaroline — Patients will have intravenous ceftaroline dosed according to current recommendations based upon its approved usage in pediatric patients for community acquired pneumonia. Blood samples will be collected for PK/PD analysis.
  Other Names: Ceftaroline fosamil,Teflaro, Zinforo

SUMMARY:
This is an open-label, single center, prospective study of patients with a diagnosis of cystic fibrosis (CF) and a history of methicillin-resistant Staphylococcus aureus (MRSA), also known as oxacillin-resistant Staphylococcus aureus (ORSA), being treated with intravenous ceftaroline. Patients will have intravenous ceftaroline dosed according to current recommendations based upon its approved usage in pediatric patients for community acquired pneumonia. The investigators will analyze pharmacokinetic (PK) and pharmacodynamic (PD) data using serum concentrations of ceftaroline measured at various time-points following infusion of ceftaroline to develop PK/PD guided dosing strategies of ceftaroline in pediatric CF patients that would be tailored to account for bacterial susceptibility and disease progression.

DETAILED DESCRIPTION:
This is an open-label, single center, prospective study of patients with a diagnosis of cystic fibrosis (CF) and a history of methicillin-resistant Staphylococcus aureus (MRSA), also known as oxacillin-resistant Staphylococcus aureus (ORSA), being treated with intravenous ceftaroline. Patients will have intravenous ceftaroline dosed according to current recommendations based upon its approved usage in pediatric patients for community acquired pneumonia. The investigators will analyze pharmacokinetic (PK) and pharmacodynamic (PD) data using serum concentrations of ceftaroline measured at various time-points following infusion of ceftaroline to develop PK/PD guided dosing strategies of ceftaroline in pediatric CF patients that would be tailored to account for bacterial susceptibility and disease progression and determine if current dosing regimes used are appropriate for this patient population.

Blood samples will be collected prior to infusion of ceftaroline and at approximately 1 hour (+/- 10 minutes), 1.5 hours (+/- 10 minutes), 3 hours (+/- 30 minutes), and 6 hours (+/- 30 minutes) after initiation of infusion. The blood samples (0.5 to 1 ml) will be collected through intravenous access, venipuncture, or capillary blood puncture. Samples will be centrifuged at 1500g at 4°C for 15 minutes within 15 minutes of collection. Serum will be separated into two aliquots of a minimum of 0.2 mL and stored at -70°C until analysis. Determination of serum ceftaroline concentrations will be measured using high-performance liquid chromatography (HPLC) method with ultraviolet (UV) detection.

Key clinical data (PK/PD) that will be collected includes age, sex, genotype, growth parameters, airway microbiology, sweat chloride values, pulmonary function test (FEV1), concomitant medications, and comorbid disorders (i.e.: CF related diabetes, CF liver disease, short gut, renal dysfunction, pulmonary hypertension, coagulopathy).

ELIGIBILITY:
Inclusion Criteria:

* Cystic Fibrosis diagnosis on accepted Cystic Fibrosis Foundation guidelines
* Inpatient
* Decision by treating physician to use intravenous ceftaroline

Exclusion Criteria:

* less than 2 years old
* 22 years of age or older
* less than 15 kg weight
* Aspartate aminotransferase (AST) or Alanine aminotransferase (ALT) > 5 fold upper limit of normal
* Gamma-glutamyltransferase (GGT) > 3 fold above upper limit of normal
* Total bilirubin > 2 mg/dL
* Platelets < 50,000
* Patients without documented CF
* Non-English speaking patients/families

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Ceftaroline Exposure and PK/PD Target Attainment | 12-hour maximum, single visit
  Interpret PK/PD target attainment based on percent time of the free ceftaroline concentration (=PK) above minimum inhibitory concentration (=PD index)

SECONDARY OUTCOMES:
FEV1 Percentage Change Assessment | 12-hour maximum, single visit
  Assess change in FEV1 percent predicted during ceftaroline treatment
Treatment Failures | 12-hour maximum, single visit
  Assess any treatment failures as evidenced by provider documentation (including FEV1 not improving and/or change in antimicrobial drugs)
Side Effects | 12-hour maximum, single visit
  Assess for side effects as documented by providers
Pulmonary Exacerbations | 12-hour maximum, single visit
  Assess for time until next pulmonary exacerbation

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Vinks, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States